CLINICAL TRIAL: NCT04827576
Title: A Phase 2, Multi-Arm Study of Magrolimab in Patients With Solid Tumors
Brief Title: Study of Magrolimab in Patients With Solid Tumors
Acronym: ELEVATELung&UC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate study
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-548-5918; 2020-005265-14 (EudraCT Number)
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — magrolimab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Run-in Cohort 1 (Magrolimab + Docetaxel) (Experimental): Participants with solid tumors (including metastatic non small cell lung cancer (mNSCLC), metastatic urothelial cancer (mUC), and metastatic small cell lung cancer (mSCLC)) will receive 1 mg/kg magrolimab intravenously (IV) on Day 1, 30 mg/kg IV on Days 8 and 15 of cycle 1; 30 mg/kg IV on Days 1, 8 and 15 of Cycle 2; 60 mg/kg IV on Day 1 of Cycle 3 and onwards for up to 113 weeks; and 75 mg/m^2 docetaxel IV on Day 1 of each cycle for up to 113 weeks; each cycle length = 21 days.
  Interventions: Drug: Magrolimab; Drug: Docetaxel
- Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) (Experimental): Participants with mNSCLC will receive 1 mg/kg magrolimab IV on Day 1, 30 mg/kg IV on Days 8 and 15 of cycle 1; 30 mg/kg IV on Days 1, 8 and 15 of Cycle 2; 60 mg/kg IV on Day 1 of Cycle 3 and onwards for up to 90 weeks; and 75 mg/m^2 docetaxel IV on Day 1 of each cycle for up to 69 weeks; each cycle length = 21 days.
  Interventions: Drug: Magrolimab; Drug: Docetaxel
- Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) (Experimental): Participants with mUC will receive 1 mg/kg magrolimab IV on Day 1, 30 mg/kg IV on Days 8 and 15 of cycle 1; 30 mg/kg IV on Days 1, 8 and 15 of Cycle 2; 60 mg/kg IV on Day 1 of Cycle 3 and onwards for up to 68 weeks; and 75 mg/m^2 docetaxel IV on Day 1 of each cycle for up to 68 weeks; each cycle length = 21 days.
  Interventions: Drug: Magrolimab; Drug: Docetaxel
- Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel) (Experimental): Participants with mSCLC will receive 1 mg/kg magrolimab IV on Day 1, 30 mg/kg IV on Days 8 and 15 of cycle 1; 30 mg/kg IV on Days 1, 8 and 15 of Cycle 2; 60 mg/kg IV on Day 1 of Cycle 3 and onwards for up to 72 weeks; and 75 mg/m^2 docetaxel IV on Day 1 of each cycle for up to 72 weeks; each cycle length = 21 days.
  Interventions: Drug: Magrolimab; Drug: Docetaxel

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously
  Other Names: GS-4721
Drug: Docetaxel — Administered intravenously
  Other Names: Taxotere®

SUMMARY:
The goals of this clinical study are to learn about the safety, tolerability, dosing and effectiveness of magrolimab in combination with docetaxel in participants with solid tumors.

DETAILED DESCRIPTION:
This study will consist of a Safety Run-in Cohort 1 (magrolimab + docetaxel combination). After completion of the Safety Run-in Cohort 1, Phase 2 Cohort 1 will occur as follows:

* Phase 2 Cohort 1: a cohort of participants with solid tumors (metastatic non-small cell lung cancer (mNSCLC) (Phase 2 Cohort 1a), metastatic urothelial cancer (mUC) (Phase 2 Cohort 1b), and metastatic small cell lung cancer (mSCLC) (Phase 2 Cohort 1c).

ELIGIBILITY:
Key Inclusion Criteria:

* Individual must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Adequate blood counts.
* Adequate renal function.
* Adequate liver function.
* Pretreatment blood cross-match completed.
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
* Measurable disease according to response evaluation criteria in solid tumours (RECIST) version 1.1

Cohort-Specific Inclusion Criteria:

* Safety Run-in Cohort 1: Individuals with metastatic advanced solid tumors who have had at least 1 prior line of systemic anticancer therapy (metastatic non-small cell lung cancer (mNSCLC) and metastatic small cell lung cancer (mSCLC)) in a locally advanced/metastatic setting, or 2 prior lines of systemic anticancer therapy (metastatic urothelial cancer (mUC)) in a locally advanced/metastatic setting, and not more than 3 prior lines of systemic anticancer therapy in a locally advanced/metastatic setting.
* Phase 2 Cohort 1a (mNSCLC): Individuals with NSCLC who have had treatment with platinum-based chemotherapy and immune checkpoint inhibitor therapy in a locally advanced/metastatic setting, either in combination or sequentially (unless not eligible for one of these therapies) are eligible. At least 1 prior line of systemic anticancer therapy in a locally advanced/metastatic setting is required and not more than 2 prior lines of systemic anticancer therapy in a locally advanced/metastatic setting are allowed. Individuals treated with a taxane within 12 months or individuals refractory to prior taxane treatment are excluded. Individuals whose tumors have genomic alterations are excluded.
* Phase 2 Cohort 1b (mUC): Individuals with UC who have had prior treatment with systemic chemotherapy and immune checkpoint inhibitor therapy in a locally advanced/metastatic setting (unless not eligible for one of these therapies) are eligible. At least 2 prior lines of systemic anticancer therapy in a locally advanced/metastatic setting are required and not more than 3 prior lines of systemic anticancer therapy in a locally advanced/metastatic setting are allowed. Individuals treated with a taxane within 12 months or individuals refractory to prior taxane treatment are excluded.
* Phase 2 Cohort 1c (mSCLC): Individuals with SCLC who have had prior treatment with platinum-based chemotherapy and/or immune checkpoint inhibitor therapy are eligible. At least 1 prior line of systemic anticancer therapy in a locally advanced/metastatic setting is required and not more than 2 prior lines of systemic anticancer therapy in a locally advanced/metastatic setting are allowed. Individuals treated with a taxane within 12 months or individuals refractory to prior taxane treatment are excluded.

Note: Maintenance therapies are not counted as separate lines of therapy.

Key Exclusion Criteria:

* Positive serum pregnancy test.
* Breastfeeding female.
* Active central nervous system (CNS) disease. Individuals with asymptomatic and stable, treated CNS lesions (radiation and/or surgery and/or other CNS-directed therapy who have not received corticosteroids for at least 4 weeks) are allowed.
* Red blood cell (RBC) transfusion dependence, defined as requiring more than 2 units of packed red blood cell transfusions during the 4-week period prior to screening. RBC transfusions are permitted during the screening period and prior to enrollment to meet the hemoglobin inclusion criteria.
* History of hemolytic anemia, autoimmune thrombocytopenia, or Evans syndrome in the last 3 months.
* Known hypersensitivity to any of the study drugs, the metabolites, or formulation excipient.
* Prior treatment with cluster of differentiation (CD)47 or signal regulatory protein alpha-targeting agents.
* Current participation in another interventional clinical study.
* Known inherited or acquired bleeding disorders.
* Significant disease or medical conditions, as assessed by the investigator and sponsor, that would substantially increase the risk-benefit ratio of participating in the study. This includes, but is not limited to, acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, and congestive heart failure New York Heart Association Class III-IV.
* Second malignancy, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, or other malignancies for which individuals are not on active anticancer therapies and who are in complete remission for over 3 years.
* Known active or chronic hepatitis B or C infection or human immunodeficiency virus.
* Prior anticancer therapy including but not limited to chemotherapy, immunotherapy, or investigational agents within 4 weeks prior to magrolimab is not permitted.

  * Note: Localized non-CNS radiotherapy, previous hormonal therapy with luteinizing hormone releasing hormone agonists for prostate or breast cancer, and treatment with bisphosphonates and receptor activator of nuclear factor kappa B ligand (RANKL) inhibitors are not criteria for exclusion.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (49):
- United States (21):
  - Cancer Treatment Centers of America, Goodyear, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Providence Saint John's Health Center, Santa Monica, California
  - St. Jude Hospital Yorba dba St. Joseph Heritage Healthcare, Santa Rosa, California
  - University of Miami, Deerfield Beach, Florida
  - Tallahassee Memorial Healthcare Cancer Center, Tallahassee, Florida
  - University Center and Blood Center,LLC., Athens, Georgia
  - Southeastern regional Medical Center, Newnan, Georgia
  - Saint Alphonsus Cancer Institute Caldwell, Caldwell, Idaho
  - Orchard Healthcare Research Inc, Skokie, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Virginia Piper Cancer Center (Alliant Health), Saint Paul, Minnesota
  - Comprehensive Cancer Centers of Nevada- Twain Office, Las Vegas, Nevada
  - Astera Cancer Care, East Brunswick, New Jersey
  - Oregon Health & Science University, Portland, Oregon
  - Charleston Oncology, Charleston, South Carolina
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, Dallas, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Medical Oncology Associates,PS (dba Summit Cancer Center) (includes IP Shipment), Spokane, Washington
- France (9):
  - Institut Bergonie, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Centre LÃon BÃrard Centre RÃgional de Lutte Contre Le Cancer, Lyon
  - Hopital Nord AP-HM, Marseille
  - Centre de Lutte Contre le Cancer (CLCC) - Centre Antoine Lacassagne (CAL) - Site Est, Nice
  - Hôpital de la Pitié Salpétrière, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Institut de Cancérologie de l'Ouest (ICO) - Saint-Herblain, Saint-Herblain
- Poland (3):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Wojewodzki Szpital Specjalistyczny w Siedlcach, Siedlce
- Spain (14):
  - Instituto de Investigacion Oncologica Vall de Hebron, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario de Jaen, Jaén
  - Hospital General Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital HM Sanchinarro, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Burren N, U'Ren L, Song K, Liu Y, Correa P, Tang S, et al. Biomarker analysis of magrolimab plus docetaxel in patients with 2L+ mNSCLC from ELEVATE Lung and UC, a Phase 2 multicohort study [Abstract]. J Immunother Cancer. 2024;12. doi:10.1136/jitc- 2024-SITC2024.0184.
- [Background] Van Burren N, U'Ren L, Song K, Liu Y, Correa P, Tang S, et al. Biomarker analysis of magrolimab plus docetaxel in patients with 2L+ mNSCLC from ELEVATE Lung and UC, a Phase 2 multicohort study. Poster presented at: 2024 Society for Immunotherapy of Cancer (SITC); 2024 Nov 6-10; Houston, TX, USA.
- [Background] Juan-Vidal O, Fang B, Paz-Ares LG, Ortega Granado AL, Vicuna BD, Bodnar L, et al. Magrolimab + docetaxel in previously treated patients with metastatic non-small cell lung cancer [Abstract]. J Immunother Cancer. 2024;12. doi:10.1136/jitc-2024-SITC2024.0604.
- [Background] Juan-Vidal O, Fang B, Paz-Ares LG, Ortega Granado AL, Vicuna BD, Bodnar L, et al. Magrolimab + docetaxel in previously treated patients with metastatic non-small cell lung cancer. Poster presented at: 2024 Society for Immunotherapy of Cancer (SITC); 2024 Nov 6-10; Houston, TX, USA.
- [Background] Vaishampayan UN, Puri S, Kummar S, Perez JM, Italiano A, Shao J, et al. A Phase 2 multiarm study of magrolimab in combination with docetaxel in patients with locally advanced or metastatic solid tumors: ELEVATE-Lung and UC. J Clin Oncol. 2023;41(16_suppl):TPS9142-TPS9142.
- [Background] Subbiah V, Vaishampayan UN, Puri S, Lin L, Chao M, Ramsingh G, et al. A Phase 2, multiarm study of anti-CD47 antibody, magrolimab, in combination with docetaxel in patients with locally advanced or metastatic solid tumors. J Clin Oncol. 2022;40(6_suppl):TPS584-TPS584.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-548-5918

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Spain, Poland, France, United States, and the United Kingdom.
Pre-assignment Details: 159 participants were screened.
Groups:
- Safety Run-in Cohort 1 (Magrolimab + Docetaxel); Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel): Participants with mSCLC received 1 mg/kg magrolimab IV on Day 1, 30 mg/kg IV on Days 8 and 15 of cycle 1; 30 mg/kg IV on Days 1, 8 and 15 of Cycle 2; 60 mg/kg IV on Day 1 of Cycle 3 and onwards for up to 72 weeks; and 75 mg/m^2 docetaxel IV on Day 1 of each cycle for up to 72 weeks; each cycle length = 21 days.
- Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel): Participants with mNSCLC received 1 mg/kg magrolimab IV on Day 1, 30 mg/kg IV on Days 8 and 15 of cycle 1; 30 mg/kg IV on Days 1, 8 and 15 of Cycle 2; 60 mg/kg IV on Day 1 of Cycle 3 and onwards for up to 90 weeks; and 75 mg/m^2 docetaxel IV on Day 1 of each cycle for up to 69 weeks; each cycle length = 21 days.
- Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel): Participants with mUC received 1 mg/kg magrolimab IV on Day 1, 30 mg/kg IV on Days 8 and 15 of cycle 1; 30 mg/kg IV on Days 1, 8 and 15 of Cycle 2; 60 mg/kg IV on Day 1 of Cycle 3 and onwards for up to 68 weeks; and 75 mg/m^2 docetaxel IV on Day 1 of each cycle for up to 68 weeks; each cycle length = 21 days.
Period: Overall Study
Arm/Group | Safety Run-in Cohort 1 (Magrolimab + Docetaxel) | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel)
Started | 9 | 29 | 26 | 42
Completed | 0 | 0 | 0 | 0
Not Completed | 9 | 29 | 26 | 42
Not completed — Death | 5 | 17 | 17 | 32
Not completed — Study Terminated by Sponsor | 2 | 9 | 7 | 5
Not completed — Investigator's Discretion | 1 | 0 | 2 | 5
Not completed — Withdrew Consent | 0 | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent to treat analysis set included all enrolled participants who took at least 1 dose of any study drug.
Groups:
- Safety Run-in Cohort 1 (Magrolimab + Docetaxel): Participants with solid tumors (including metastatic non small cell lung cancer (mNSCLC), metastatic urothelial cancer (mUC), and metastatic small cell lung cancer (mSCLC)) received 1 mg/kg magrolimab intravenously (IV) on Day 1, 30 mg/kg IV on Days 8 and 15 of cycle 1; 30 mg/kg IV on Days 1, 8 and 15 of Cycle 2; 60 mg/kg IV on Day 1 of Cycle 3 and onwards for up to 113 weeks; and 75 mg/m^2 docetaxel IV on Day 1 of each cycle for up to 113 weeks; each cycle length = 21 days.
Arm/Group | Safety Run-in Cohort 1 (Magrolimab + Docetaxel) | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel) | Total~(N=106)
Number analyzed (Participants) | 9 | 29 | 26 | 42 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 13 | 12 | 27 | 57
  >=65 years | 4 | 16 | 14 | 15 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8.2) | 63 (10.8) | 65 (9.8) | 62 (6.6) | 63 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 7 | 17 | 34
  Male | 5 | 23 | 19 | 25 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 1 | 4
  Not Hispanic or Latino | 8 | 25 | 20 | 30 | 83
  Unknown or Not Reported | 1 | 1 | 6 | 11 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 2
  White | 7 | 27 | 19 | 30 | 83
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 6 | 11 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 0 | 17 | 9 | 14 | 40
  United States | 9 | 9 | 9 | 12 | 39
  France | 0 | 1 | 6 | 11 | 18
  Poland | 0 | 2 | 0 | 4 | 6
  United Kingdom | 0 | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any adverse events (AE) not present prior to the study treatment, or any events already present but worsening in either intensity or frequency following exposure to the study treatment. The TEAE reporting period is defined as the period from the date of the first dose of study treatment up to 30 days after the date of the last dose of study treatment or the day before initiation of subsequent antineoplastic therapy, whichever comes first. An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution.
Time Frame: First dose date up to 113 weeks plus 30 days
Population: Participants in the Safety Analysis Set were analyzed. The Safety Analysis Set included all participants who took at least 1 dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Safety Run-in Cohort 1 (Magrolimab + Docetaxel) | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel)
Number analyzed (Participants) | 9 | 29 | 26 | 42
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days and prior to the day of initiation of subsequent anti-cancer therapy. Percentages were rounded off.
Time Frame: First dose date up to 113 weeks plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Safety Run-in Cohort 1 (Magrolimab + Docetaxel) | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel)
Number analyzed (Participants) | 9 | 29 | 26 | 42
percentage of participants
  Any Grade | 100 | 100 | 100 | 100
  Grade 3 or Higher | 77.8 | 82.8 | 92.3 | 78.6

3. Primary Outcome: Objective Response Rate (ORR) (Phase 2 Cohorts 1a, 1b, and 1c)
Description: ORR was defined as the percentage of participants who achieved a complete response (CR) or partial response (PR), as measured by RECIST version 1.1, as determined by investigator assessment. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Clopper-Pearson method was used in outcome measure analysis. Percentages were rounded-off.
Time Frame: Up to 90 Weeks
Population: Participants in the modified intent to treat analysis set were analyzed. The study had 2 parts - Safety Run-in and Phase 2. Per pre-specified analysis, this endpoint was applicable only to Phase 2 cohorts. Therefore, data for cohorts of Phase 2 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel)
Number analyzed (Participants) | 29 | 26 | 42
percentage of participants | 17.2 [5.8 to 35.8] | 3.8 [0.1 to 19.6] | 4.8 [0.6 to 16.2]

4. Secondary Outcome: Progression-free Survival (PFS) (Phase 2 Cohorts 1a, 1b, and 1c)
Description: PFS was defined as the interval from the first dosing date of any study drug to the earlier date of the first documentation of objective disease progression (PD) by investigator assessment per RECIST, Version 1.1, or death from any cause. PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (the appearance of one or more new lesions was also considered progression). Kaplan-Meier (KM) estimates were used in outcome measure analysis.
Time Frame: Up to 117 Weeks
Population: Participants in the modified Intent-to-Treat Analysis Set were analyzed. The study had 2 parts - Safety Run-in and Phase 2. Per pre-specified analysis, this endpoint was applicable only to Phase 2 cohorts. Therefore, data for cohorts of Phase 2 are reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel)
Number analyzed (Participants) | 29 | 26 | 42
months | 4.2 [2.0 to 8.0] | 2.7 [2.1 to 4.0] | 2.2 [2.0 to 3.9]

5. Secondary Outcome: Duration of Response (DOR) (Phase 2 Cohorts 1a, 1b, and 1c)
Description: DOR was defined as time from first documentation of CR or PR to the earliest date of documented PD, per RECIST, Version 1.1, or death from any cause, whichever occurs first, as determined by investigator assessment. CR and PR are defined in outcome measure #3 and PD is defined in outcome measure #4. KM Estimates were used in outcome measure analysis.
Time Frame: Up to 117 Weeks
Population: Participants in the modified Intent-to-Treat Analysis Set who achieved CR or PR were analyzed. The study had 2 parts - Safety Run-in and Phase 2. Per pre-specified analysis, this endpoint was applicable only to Phase 2 cohorts. Therefore, data for cohorts of Phase 2 are reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel)
Number analyzed (Participants) | 5 | 1 | 2
months | 7.6 [3.7 to NA] — Upper limit of confidence interval was not estimable due to low number of participants with events. | NA [NA to NA] — Median, lower and upper limit of confidence interval were not estimable due to low number of participants with events. | 4.7 [4.6 to NA] — Upper limit of confidence interval was not estimable due to low number of participants with events.

6. Secondary Outcome: Overall Survival (OS) (Phase 2 Cohorts 1a, 1b, and 1c)
Description: OS is defined as time from date of dose initiation to death from any cause. KM estimates were used in outcome measure analysis.
Time Frame: Up to 117 Weeks
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel)
Number analyzed (Participants) | 29 | 26 | 42
months | 9.8 [5.2 to NA] — Upper limit of confidence interval was not estimable due to low number of participants with events. | 7.6 [4.7 to 13.7] | 6.4 [3.9 to 8.3]

7. Secondary Outcome: Serum Concentration of Magrolimab
Time Frame: Day 1, Day 8 Predose, Day 8 1-Hour Postdose, Day 22, Day 43 Predose, Day 43 1-Hour Postdose, Day 85, Day 127, Day 190 and Day 253 Predose
Population: The participants in the Pharmacokinetic (PK) Analysis Set with available data were analyzed. The PK Analysis Set included all participants who received any amount of magrolimab and have at least 1 measurable posttreatment serum concentration of magrolimab. Here 'N' is defined as participants with available data at the given timepoint.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Safety Run-in Cohort 1 (Magrolimab + Docetaxel) | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel)
Number analyzed (Participants) | 7 | 23 | 23 | 36
μg/mL
  Day 1 Predose | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Day 8 Predose: number analyzed (Participants) | 5 | 20 | 22 | 29
  Day 8 Predose | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Day 8 1-Hour Postdose: number analyzed (Participants) | 1 | 0 | 0 | 0
  Day 8 1-Hour Postdose | 407 (NA) — Standard Deviation (SD) is not estimable for 1 participant. |  |  |
  Day 22 Predose: number analyzed (Participants) | 4 | 23 | 23 | 32
  Day 22 Predose | 460 (112) | 302 (161) | 260 (148) | 334 (134)
  Day 43 Predose: number analyzed (Participants) | 5 | 20 | 21 | 28
  Day 43 Predose | 624 (451) | 523 (195) | 439 (182) | 529 (258)
  Day 43 1- Hour Postdose: number analyzed (Participants) | 2 | 18 | 18 | 27
  Day 43 1- Hour Postdose | 1880 (523) | 1550 (525) | 1560 (492) | 1730 (560)
  Day 85 Predose: number analyzed (Participants) | 4 | 14 | 12 | 15
  Day 85 Predose | 415 (135) | 266 (134) | 319 (271) | 297 (181)
  Day 127 Predose: number analyzed (Participants) | 3 | 11 | 3 | 10
  Day 127 Predose | 277 (35.0) | 281 (143) | 393 (93.8) | 174 (106)
  Day 190 Predose: number analyzed (Participants) | 3 | 7 | 0 | 4
  Day 190 Predose | 281 (71.1) | 344 (104) |  | 250 (113)
  Day 253 Predose: number analyzed (Participants) | 2 | 6 | 0 | 0
  Day 253 Predose | 237 (56.6) | 363 (179) |  |

8. Secondary Outcome: Percentage of Participants Who Developed Anti-Magrolimab Antibodies
Time Frame: Up to 113 Weeks
Population: Participants in the Immunogenicity Analysis Set with available data were analyzed. The Immunogenicity Analysis Set includes all participants who received any amount of magrolimab and have at least 1 evaluable anti-magrolimab antibody test result.
Measure: Number; unit: percentage of participants
Arm/Group | Safety Run-in Cohort 1 (Magrolimab + Docetaxel) | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel)
Number analyzed (Participants) | 7 | 25 | 25 | 37
percentage of participants | 0 | 4.0 | 8.0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 117 weeks; Adverse events: Up to 113 weeks plus 30 days
Description: All-cause mortality: All Enrolled Analysis Set included all participants who received a study subject identification number in the study after screening. Adverse events: The Safety Analysis Set included all participants who took at least 1 dose of any study drug.
Arm/Group | Safety Run-in Cohort 1 (Magrolimab + Docetaxel) | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel)
All-Cause Mortality (participants affected / at risk) | 6/9 | 17/29 | 18/26 | 37/42
Serious Adverse Events (participants affected / at risk) | 5/9 | 16/29 | 12/26 | 18/42
Other Adverse Events (participants affected / at risk) | 9/9 | 29/29 | 26/26 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Cohort 1 (Magrolimab + Docetaxel) (N=9) | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) (N=29) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) (N=26) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel) (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 4 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 4 | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1
Neuritis (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Cohort 1 (Magrolimab + Docetaxel) (N=9) | Phase 2 Cohort 1a, mNSCLC (Magrolimab + Docetaxel) (N=29) | Phase 2 Cohort 1b, mUC (Magrolimab + Docetaxel) (N=26) | Phase 2 Cohort 1c, mSCLC (Magrolimab + Docetaxel) (N=42)
Anaemia (Blood and lymphatic system disorders) | 5 | 22 | 14 | 26
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 5 | 4 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 13 | 13 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 5 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 6 | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 2 | 14 | 6 | 19
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 5 | 4 | 16
Stomatitis (Gastrointestinal disorders) | 0 | 4 | 3 | 5
Vomiting (Gastrointestinal disorders) | 2 | 4 | 4 | 7
Asthenia (General disorders) | 1 | 18 | 10 | 23
Chills (General disorders) | 1 | 0 | 1 | 4
Fatigue (General disorders) | 6 | 6 | 5 | 11
Generalised oedema (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 3 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 2 | 2
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 3 | 6 | 5 | 4
Pyrexia (General disorders) | 3 | 11 | 8 | 8
Vascular device occlusion (General disorders) | 1 | 0 | 0 | 0
Contrast media reaction (Immune system disorders) | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 1 | 3
Covid-19 (Infections and infestations) | 0 | 2 | 1 | 1
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Nail infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 2 | 0 | 1 | 3
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 4
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 4 | 2
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 4 | 2 | 5
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 3
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 2
C-reactive protein increased (Investigations) | 0 | 0 | 2 | 1
Lymphocyte count decreased (Investigations) | 2 | 3 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 4 | 0 | 3
Sars-cov-2 test positive (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 2 | 3
White blood cell count decreased (Investigations) | 2 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7 | 2 | 17
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 5 | 1 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 2
Iron overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 4
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 6
Dysgeusia (Nervous system disorders) | 1 | 2 | 2 | 6
Headache (Nervous system disorders) | 2 | 1 | 2 | 6
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 6 | 1 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 3
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 2
Depression (Psychiatric disorders) | 3 | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 2 | 3
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 3 | 12
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 8 | 6 | 6
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 0
Hypotension (Vascular disorders) | 1 | 3 | 0 | 2
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT04827576/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-06): https://cdn.clinicaltrials.gov/large-docs/76/NCT04827576/SAP_001.pdf